CLINICAL TRIAL: NCT06178744
Title: Outcome Reflection for Immune Mediated Rejection by Utilizing Artificial Intelligence in Cardiac Transplant Patients Through Early and Late Echocardiographic Analysis (ORACLE)
Brief Title: A Study of AI in Cardiac Transplant in Echocardiographic Analysis (ORACLE)
Acronym: ORACLE
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Atta Behfar MD, PhD, Principal Investigator, Mayo Clinic
Other Study IDs: 23-006378
Record Dates: First submitted 2023-12-12; First posted 2023-12-21 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this research is to detect episodes of rejection versus non-rejection after cardiac transplant and the diagnostic accuracy of an Artificial Intelligence (AI) algorithm using the data from an ECG (electrocardiogram) and Cardiac Ultrasound (Echocardiogram and/or point of care ultrasound).

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing post-cardiac transplant endomyocardial biopsy, and the ability to provide informed consent and a consent for the study.

Exclusion Criteria:

* Refusal of study participation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Post-cardiac transplantation subjects, presenting to the cardiac catheterization laboratories at Mayo Clinic in Rochester, MN for routine surveillance biopsies or for diagnostic biopsies in the setting of clinical concern including rejection and graft dysfunction will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Number of episodes identified by the Artificial Intelligence (AI) algorithm as 1R or greater acute cellular rejection, grade 1 or greater antibody mediated rejection, reduction in LVEF to <50%, or a drop in LVEF >5% | 2 years
  Number of episodes identified by the AI algorithm as 1R or greater acute cellular rejection, grade 1 or greater antibody mediated rejection, reduction in LVEF to <50%, or a drop in LVEF >5% utilizing electrocardiograms and cardiac ultrasound images/videos obtained from point of care ultrasound (POCUS) or echocardiograms.

CONTACTS AND LOCATIONS:
Overall Officials: Atta Behfar, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No